CLINICAL TRIAL: NCT03414801
Title: A Single-Group Study Evaluating Reproducibility of Rhinitis Symptoms Induced by Cat Allergen (Fel d1) Exposure in the Red Maple Trials Natural Exposure Chamber (NEC) ™ in Subjects With Cat Allergy
Brief Title: Red Maple Trials Cat Allergen Natural Exposure Chamber Validation in Cat-allergic Subjects
Acronym: NEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Red Maple Trials Inc. (Industry)
Collaborators: Ottawa Allergy Research Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RMT005
Record Dates: First submitted 2018-01-18; First posted 2018-01-30 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-04

CONDITIONS: Allergic Rhinitis; Rhinoconjunctivitis; Exposure
Keywords: Environmental Exposure Unit; Cat Allergen; Rhinitis; Subject Validation
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis | interventions — Environmental Exposure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Active Comparator): Cat Allergic Subjects
  Interventions: Other: Allergen Exposure
- Cohort 2 (Active Comparator): Non-Allergic Subjects will
  Interventions: Other: Allergen Exposure

INTERVENTIONS:
Other: Allergen Exposure — Subjects will undergo two exposure sessions, one week apart, of up to 1 hour depending on the subject's symptom severity and pulmonary function. During the exposure, subjects will be exposed to cat dander and levels of cat allergen, Fel d1, will be measured using sampling pumps with attached filters.
  Other Names: Environmental Exposure

SUMMARY:
To assess the reproducibility of the allergic response in the cat allergic subjects, measured as the change from baseline of the Total Nasal Symptom Score (TNSS) on the two challenge days.

DETAILED DESCRIPTION:
To validate the Red Maple Trials Natural Exposure Chamber for cat exposure studies in non-asthmatic subjects with perennial allergic rhinitis and allergy to cat dander by examining the reproducibility of the response on two allergen challenge days and comparing the response of allergic to non-allergic subjects.

ELIGIBILITY:
Inclusion Criteria for Allergic Subjects:

* Male and female adults, 18 years to 65 years of age
* Willing and able to give informed consent for participation in the study.
* Otherwise healthy with a diagnosis of perennial allergic rhinitis and a clinical history of nasal symptoms during exposure to cat in the previous 2 years
* With positive skin prick test reactivity to cat dander. A positive skin prick test is a wheal ≥3 mm larger than the negative control performed at the screening visit or within 6 months of the screening visit provided that complete documentation (specific allergen used for the SPT and the size of the reaction) is available
* Having sufficient rhinoconjunctivitis symptoms (TRCSS score ≥5) during the first cat challenge
* If subjects are taking medications (other than allergy medications), the dosing must be stable for at least 4 weeks prior to study entry
* With laboratory results at the screening visit which, in the opinion of the investigator, are clinically acceptable for the subject to be enrolled in the study
* Able (in the investigators opinion) and willing to comply with all study requirements

Exclusion Criteria for Allergic Subjects:

* Subjects with a cat at home or who are regularly exposed to cats during the study period
* Subjects with a diagnosis of asthma with the exception of mild intermittent asthma defined as normal lung function and intermittent treatment with a short-acting beta agonist only
* Subjects with a history of anaphylactic reactions defined as previous or current presentation with two or more of the following:

  * Involvement of the skin or mucosa
  * respiratory difficulties
  * low blood pressure
  * gastrointestinal symptoms
* Subjects who have undergone allergen desensitization for cat allergy within the last 2 years
* Subjects with structural nasal defects or nasal polyps
* Subjects with a positive skin-prick test reaction to house dust mite
* Subjects having an infection of the upper airways within 2 weeks prior to the screening visit.
* Subjects who develop an upper respiratory tract infection during the study will be discontinued
* Subjects who have received treatment with Xolair or immunosuppressants during the 4 months prior to the screening visit
* Subjects who wear contact lenses will not be permitted to wear them during the challenge sessions
* Female subjects who are pregnant or lactating at screening or who are planning pregnancy during the course of the study
* Subjects with significant renal or hepatic impairment at screening
* Subjects with scheduled elective surgery or other procedures requiring general anaesthesia during the study
* Subjects with any other significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the outcomes of the study, or the participant's ability to participate in the study
* Subjects who have participated in another research study involving an investigational product within 30 days or 5 half-lives prior to the screening visit
* Subjects who are using unacceptable concomitant medications within the washout period prior to the screening visit (see Table 7.2-1)
* Subjects with a history of alcohol or drug abuse within the previous 5 years
* Subjects with known HIV or hepatitis B or C positivity
* Subjects who for any reason would be unlikely to comply with the study requirements

Inclusion Criteria for non allergic subjects:

* Healthy male and female adults, 18 years to 65 years of age
* Willing and able to give informed consent for participation in the study.
* With laboratory results at the screening visit which, in the opinion of the investigator, are clinically acceptable for the subject to be enrolled in the study
* Able (in the investigators opinion) and willing to comply with all study requirements

Exclusion Criteria for non allergic subjects:

* With a diagnosis of perennial allergic rhinitis and a clinical history of nasal symptoms during exposure to cat in the previous 2 years
* With positive skin prick test reactivity to cat dander. A positive skin prick test is a wheal ≥3 mm larger than the negative control performed at the screening visit
* Subjects with a cat at home or who are regularly exposed to cats during the study period
* Subjects with a diagnosis of asthma with the exception of mild intermittent asthma defined as normal lung function and intermittent treatment with a short-acting beta agonist only
* Subjects with a history of anaphylactic reactions defined as previous or current presentation with two or more of the following:

  * Involvement of the skin or mucosa
  * respiratory difficulties
  * low blood pressure
  * gastrointestinal symptoms
* Subjects with structural nasal defects or nasal polyps
* Subjects with a positive skin-prick test reaction to house dust mite
* Subjects having an infection of the upper airways within 2 weeks prior to the screening visit.
* Subjects who develop an upper respiratory tract infection during the study will be discontinued
* Subjects who have received treatment with Xolair or immunosuppressants during the 4 months prior to the screening visit
* Subjects who wear contact lenses will not be permitted to wear them during the challenge sessions
* Female subjects who are pregnant or lactating at screening or who are planning pregnancy during the course of the study
* Subjects with significant renal or hepatic impairment at screening
* Subjects with scheduled elective surgery or other procedures requiring general anaesthesia during the study
* Subjects with any other significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the outcomes of the study, or the participant's ability to participate in the study
* Subjects who have participated in another research study involving an investigational product within 30 days or 5 half-lives prior to the screening visit
* Subjects who are using unacceptable concomitant medications within the washout period prior to the screening visit (see Table 7.2-1)
* Subjects with a history of alcohol or drug abuse within the previous 5 years
* Subjects with known HIV or hepatitis B or C positivity
* Subjects who for any reason would be unlikely to comply with the study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Difference in Total Nasal Symptom Score (TNSS) change from baseline to the end of the challenge between the two challenge days (Visits 2 and 3) in the cat-allergic subjects | 15 weeks
  Runny nose, sneezing, blocked nose, itchy nose

SECONDARY OUTCOMES:
TNSS change from baseline to the end of the challenge of allergic subjects to non-allergic subjects | 15 weeks
Difference in exposure time between the two exposure days for all subjects | 15 weeks
Comparison of the exposure times of allergic compared to non-allergic subjects | 15 weeks
Comparison of TNSS at individual time points on the two exposure days | 15 weeks
  Runny nose, sneezing, blocked nose, itchy nose
Comparison of Total Respiratory Symptom Score (TRSS) at individual time points on the two exposure days | 15 weeks
  Wheezing, shortness of breath, coughing
Comparison of Total Rhinoconjunctivitis Symptom Score (TRCSS) at individual time points on the two exposure days | 15 weeks
  Sum of TNSS and TOSS
Comparison of Total Ocular Symptom Score (TOSS) at individual time points on the two exposure days | 15 weeks
  Itchy eyes and watery eyes
Comparison of Fel d1 levels during the exposures | 15 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ottawa Allergy Research Corporation, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No